CLINICAL TRIAL: NCT00962611
Title: An Open Label Phase I Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Maximum Tolerated Dose and Biomarker Response After Intravenous Administration of Weekly BAY80-6946 to Patients With Advanced Cancer
Brief Title: BAY80-6946 Open Label, Phase I Study in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12871
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: Solid tumors; Advanced cancer
MeSH Terms: conditions — Neoplasms | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Copanlisib (Experimental)
  Interventions: Drug: Copanlisib (Aliqopa, BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (Aliqopa, BAY80-6946) — BAY80-6946 given IV over 1 hour every week for three weeks with a one week break until progression or unacceptable toxicities develop.

SUMMARY:
The purpose of this study is to determine the tolerability, maximum tolerated dose and pharmacokinetics of this drug.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years.
* Histological or cytological documentation of non-hematologic, malignant solid tumor, excluding primary brain or spinal tumors, or history of central nervous system metastases
* At least one measurable lesion or evaluable disease
* Life expectancy of at least 12 weeks
* ECOG Performance Status of 0, 1 or 2
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists]. Low-dose aspirin is permitted (</= 100 mg daily).
* Adequate bone marrow, liver and renal function
* Ability to understand and to sign an informed consent form; a signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* History of cardiac disease congestive heart failure (CHF) > NYHA Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months prior to study entry or unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or Digoxin are permitted).
* Current diagnosis of type I or II diabetes mellitus or fasting blood glucose level >125 mg/dL at screening, or HbA1c 7%
* Active clinically serious infections > Grade 2 (NCI-CTCAE Version 3.0)
* History of having received allogeneic organ transplant
* Uncontrolled seizure disorder. Use of cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital) is not allowed throughout the entire study.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-11-19 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
Characterize safety, tolerability + pharmacokinetics, to determine the maximum tolerated dose of BAY80-6946 administered 1x weekly for 3 weeks, every 4weeks, as a 1h-intravenous infusion. Evaluate biomarkers that may be predictive of tumor response. | 2 years

SECONDARY OUTCOMES:
Determine the effects of BAY80-6946 on blood glucose and insulin, and its safety in patients with type I or II diabetes. | 2 years
Evaluate for early signs of efficacy in expansion cohorts | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - Pittsburgh, Pennsylvania
  - San Antonio, Texas

REFERENCES:
- [Background] A. Patnaik et al. Supplementary materials /Supplementary methods. Annals of Oncology 2016
- [Result] Rowe EL. Automated drop volume apparatus for surface tension measurement. J Pharm Sci. 1972 May;61(5):781-2. doi: 10.1002/jps.2600610523. No abstract available. PMID 5035790
- [Derived] Patnaik A, Appleman LJ, Tolcher AW, Papadopoulos KP, Beeram M, Rasco DW, Weiss GJ, Sachdev JC, Chadha M, Fulk M, Ejadi S, Mountz JM, Lotze MT, Toledo FG, Chu E, Jeffers M, Pena C, Xia C, Reif S, Genvresse I, Ramanathan RK. First-in-human phase I study of copanlisib (BAY 80-6946), an intravenous pan-class I phosphatidylinositol 3-kinase inhibitor, in patients with advanced solid tumors and non-Hodgkin's lymphomas. Ann Oncol. 2016 Oct;27(10):1928-40. doi: 10.1093/annonc/mdw282. PMID 27672108